CLINICAL TRIAL: NCT03924219
Title: Assessment of CMV-specific T Cell Responses by Flow Cytometry With Intracellular Cytokine Staining to Predict CMV Infection Risk in Pediatric Solid Organ Transplant Recipients
Brief Title: CMV T Cell Immunity in Pediatric Solid Organ Transplant Recipients
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: ViraCor Laboratories (Industry)
Responsible Party: Principal Investigator, Daniel Dulek, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 180947
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplant Infection; Kidney Transplant Infection; Liver Transplant Infection; CMV
Keywords: cmv
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Solid Organ Transplant (SOT) Recipients: Pediatric patients (<18 years of age) undergoing or anticipated to undergo solid organ transplantation (heart, kidney, or liver) will be prospectively enrolled with serial blood collection for CMV T cell Immunity Assay performance.
  Interventions: Other: CMV T cell Immunity Assay

INTERVENTIONS:
Other: CMV T cell Immunity Assay — Flow cytometry based assay quantifying IFN-gamma expression in T cells following CMV peptide stimulation (Viracor)

SUMMARY:
CMV infection and disease remain a significant clinical challenge for pediatric solid organ transplant (SOT) recipients. Current prevention strategies are limited to prophylaxis in which antiviral medication is administered for a period of several months or preemption in which close monitoring of CMV viral load from the peripheral blood is performed and treatment is initiated when CMV is detected. Each of these strategies has risks, costs, and limitations associated with it. Recently, assays for measurement of an individual patient's CMV immunity have been developed and are clinically available. One of these is the Viracor CMV T cell Immunity Panel. This flow cytometry based assay is performed on peripheral blood and measures cytokine release in response to CMV antigen stimulation by flow cytometry. The thresholds for this assay that confer protection against CMV infection in pediatric SOT recipients are not known. Defining CMV-specific cell mediated immune response thresholds that confer protection against CMV reactivation could inform patient specific durations of antiviral prophylaxis or pre-emptive surveillance testing. Therefore, the objective of this study is to quantify CMVresponsive T lymphocyte populations by flow cytometry (Viracor CMV T cell Immunity Panel) in pediatric heart, kidney, and liver transplant recipients within the first year of transplantation and to investigate potential threshold values that correlate with protection against CMV infection (DNAemia).

ELIGIBILITY:
Inclusion Criteria:

1. < 18 years of age at the time of pre-transplant enrollment
2. Potential subject is undergoing evaluation or is currently listed for isolated heart, kidney, or liver transplantation at a participating transplant center OR is anticipated to undergo living-donor kidney or liver transplantation
3. Anticipated to receive ≤ 200 days of antiviral chemoprophylaxis

Note: Subjects who are consented, enrolled, and undergo transplantation at <18 years of age will remain in the study and be followed post-transplant according to the study plan after they turn 18 years of age. Subjects will be re-consented to remain in the study at their first study visit after turning 18 years of age.

Exclusion Criteria:

I. Exclusion Criteria pre-transplant

1. Prior history of any organ transplant
2. Prior history of hematopoietic cell transplant
3. Anticipated to receive more than one organ at the time of transplant
4. Anticipated to receive > 200 days of CMV antiviral chemoprophylaxis as part of the local transplant center's standard CMV prevention protocol
5. History of underlying primary (genetic) T cell immune deficiency

II. Exclusion Criteria post-enrollment A) Removal from study due to minimal risk for CMV infection

1. CMV seronegative children >= 12 months of age will be enrolled pre-transplant but will subsequently be excluded from the study IF they receive an organ from a CMV seronegative donor (CMV D-/R-).
2. Infants <12 months will be considered seronegative regardless of their CMV IgG status (whether or not this testing was obtained by the local transplant center) UNLESS the infant has a positive pre-transplant CMV culture (from urine) or a positive pre-transplant CMV PCR (from urine, saliva, or blood). Infants <12 months of age without evidence of prior CMV infection (as defined by these preceding criteria) will be excluded from post-transplant follow up IF they receive an organ from a CMV seronegative donor due to low risk for post-transplant CMV infection. Infants <12 months of age with evidence of prior CMV infection (as defined above) will remain in the study following transplantation.

B) Removal from study due to age

a. Subjects who are enrolled at <18 years of age but are not transplanted prior to their 18th birthday will be removed from the study and will not have further pre- or post-transplant follow up.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients <18 years of age listed or anticipated to undergo kidney, heart, or liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
CMV Infection Incidence | 12 months post-transplantation
  CMV Infection as measured by CMV DNAemia or CMV disease

SECONDARY OUTCOMES:
Frequency of detectable CMV T cell Immunity | 12 months post-transplantation
  Viracor T cell Immunity Assay

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dulek, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (12):
- United States (12):
  - Stanford University Medical Center/Lucile Packard Children's Hospital Stanford, Stanford, California
  - Emory University Medical Center/Children's Hospital of Atlanta, Atlanta, Georgia
  - Northwestern University Medical Center/Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albert Einstein College of Medicine/Children's Hospital at Montefiore, New York, New York
  - Duke University Medical Center/Duke Children's Hosptial, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center/Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No